CLINICAL TRIAL: NCT04087681
Title: Pilot Study to Assess Success Factors and Barriers for Preparation of a Phase 3 Study With ExPEC10V in Adults Aged 60 Years or Older and in Stable Health
Brief Title: Study to Collect Information About Invasive Disease Caused by Extraintestinal Pathogenic Escherichia Coli (EXPECT-1)
Acronym: EXPECT-1
Status: Completed | Type: Observational
Sponsor: MJM Bonten (Other)
Collaborators: Janssen Research & Development, LLC (Industry); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor-Investigator, MJM Bonten, Professor doctor, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: VAC52416BAC0005
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: E.Coli Infections
Keywords: Extraintestinal pathogenic Escherichia coli (ExPEC); Invasive ExPEC disease (IED); Pilot study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly 60+ preferably those with increased risk of IED: Study participants are aged 60 years or older in stable health, preferably with a history of urinary tract infection in the previous 10 years.

SUMMARY:
The purpose of this study is to collect information from study participants who develop an invasive disease caused by Extraintestinal pathogenic E. coli (ExPEC) during a period of 12 months. This information will be used to support the development of a new vaccine to prevent ExPEC infections.

DETAILED DESCRIPTION:
Invasive ExPEC disease (IED) is defined as an acute illness consistent with bacterial infection that is microbiologically confirmed by the isolation and identification of E. coli from blood or other normally sterile body sites, or by the isolation and identification of E. coli from urine in a patient with signs and symptoms of invasive disease and no other identifiable source of infection. Adults aged 60 years or older have an increased risk of developing IED. To date, there is no vaccine available to prevent IED. ExPEC10V is a 10 valent vaccine candidate in development by Janssen R&D for the prevention of IED in adults aged 60 years and older. A Phase 3 clinical study is planned to investigate the efficacy and safety of this vaccine. To obtain insight in the feasibility and design of the Phase 3 study, a pilot study is required.

This pilot study is a prospective, multicenter, observational study conducted in a maximum of eight countries in Europe, North-America and Asia. Participant recruitment will be done in primary care. In each participating country a local primary care network encompassing approximately 40,000 persons and a local hospital, where patients are referred to in case of a suspicion of IED, will participate in this study.

Database screening at the primary care centers will be performed to identify and invite potential eligible study participants. Upon consent, each study participant will be followed for a period of maximum 12 months after enrollment in the study. At baseline, demographic data and medical history data will be collected. During the follow-up period, any referral of study participants to a hospital for any reason including IED will be collected. IED identification and Medical Resource Utilization (MRU) during the follow-up period will be performed by regular telephone calls with all study participants. At the end of the study, the primary care files will also be checked for MRU. If a participant is diagnosed with IED and admitted to the hospital, the following data will be collected: medical history and treatment received 90 days prior to the IED, clinical and laboratory data, data on the treatment and outcome of IED and data on MRU related to IED. Data will be collected on Day 1 of IED diagnosis (signs/ symptoms) and Day 28 after IED diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing to provide written informed consent prior to inclusion.
* Participant is male or female preferably with a history of UTI in the previous 10 years. Participant without a (known) history of UTI in the previous ten years may also be enrolled.
* Participant is aged 60 years or older on the day of signing the informed consent form (ICF).
* Participant is willing to be available for contact with investigator for the duration of the study.
* Participant is ambulatory and lives in the community or in assisted-living or long-term care residential facility that provides minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.
* Based on the clinical judgment of the investigator, participant must be in stable health. Participants may have underlying illnesses such as hypertension, congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD), type 2 diabetes mellitus, as long as their signs and symptoms are stable and medically controlled.

Exclusion Criteria:

* Participant has a serious chronic disorder, including severe COPD or clinically significant CHF, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, Alzheimer's disease, or has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g. compromise well-being) or that could prevent, limit, or confound the protocol-specified assessments.
* Participant has history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence).
* Participant has had major psychiatric illness and/or drug or alcohol abuse which in investigators opinion would compromise the participant's safety and/or compliance with the study procedures.
* Participant who, in the opinion of the investigator, is unlikely to adhere to the requirements of the study, or is unlikely to complete the full course of the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes male and female participants aged 60 years or older in stable health, preferably at increased risk for IED. A total of 6,000 study participants will be recruited. At least 50% of the study participants will be healthy elderly aged 60 years or older with a history of UTI in the previous ten years. The other 50% of participants will be healthy elderly aged 60 years or older with no (known) history of UTI in the previous ten years.
Sampling Method: Non-Probability Sample
Enrollment: 4479 (Actual)
Dates: Start 2019-09-28 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Participant enrolment rate (% of patients screened/invited vs. enrolled) | 3 months
  Participant enrolment rate (% of patients screened/invited vs. enrolled)
Number of hospital admissions of participants reported by the hospital versus the number of hospital admissions obtained through medical record checks by the primary care center versus the number of hospital admissions reported by participants narrative | 12 months
  Number of hospital admissions of participants reported by the hospital versus the number of hospital admissions obtained through medical record checks by the primary care center versus the number of hospital admissions reported by participants narrative
Number of IED hospital admissions of participants reported by the hospital vs. the number of IED hospital admissions obtained by medical record checks of the primary care center vs. the number of IED hospital admissions reported by participants narrative | 12 months
  Number of IED hospital admissions of participants reported by the hospital vs. the number of IED hospital admissions obtained by medical record checks of the primary care center vs. the number of IED hospital admissions reported by participants narrative
Description of medical assessment pathways based on participants medical files. | 12 months
  Description of medical assessment pathways based on participants medical
Description of standard of care diagnostic methods based on participants medical files. | 12 months
  Description of standard of care diagnostic methods based on participants medical files.
Description of treatment of bacteremic and nonbacteremic IED based on participants medical files. | 12 months
  Description of treatment of bacteremic and nonbacteremic IED based on participants medical files.
Incidence of IED (number % of IED cases in the group of study participants) | 12 months
  Incidence of IED (number % of IED cases in the group of study participants)

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Ekkelenkamp, Dr., Principal Investigator — UMC Utrecht
Locations (8):
- Duke Clinical Research Institute, Durham, North Carolina, United States
- Duke Clinical Research Institute, Greater Sudbury, Canada
- Chu Limoges - Cic, Limoges, France
- UKK Uniclinic Cologne, Cologne, Germany
- University of Verona, Verona, Italy
- Janssen Pharmaceutical K.K., Tokyo, Chiyoda-ku, Japan
- - Andalusian Public Foundation for Health Research Management in Seville (FISEVI), Seville, Spain
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No